CLINICAL TRIAL: NCT01794286
Title: Improving Childhood Immunization Compliance Using Electronic Health Records
Brief Title: Improving Childhood Immunization
Acronym: ImmProve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Marlene Miller, Professor, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RC1LM010512 (NIH)
Record Dates: First submitted 2013-02-13; First posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Improve Childhood Immunization Rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Trigger alerts only
  Interventions: Other: Trigger alerts
- Intervention Group (Experimental): Trigger alerts + provider bulletins
  Interventions: Other: Provider bulletins; Other: Trigger alerts

INTERVENTIONS:
Other: Provider bulletins
  Arms: Intervention Group
Other: Trigger alerts

SUMMARY:
Specific Aim: To improve childhood immunization rates by utilizing automated Electronic Health Record-derived provider-specific performance feedback reports, coupled with automated Electronic Health Record-derived trigger alerts.

Hypothesis: The automated Electronic Health Record-derived provider-specific performance feedback reports will result in a 50% decrease in unimmunized children ages 0-13 years of age, when coupled with automated Electronic Health Record-derived trigger alerts, compared with trigger alerts alone.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric resident providers in Harriet Lane Clinic at Johns Hopkins University

Exclusion Criteria:

* none

Ages: 28 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Receipt of missing immunization | Time to event analyses, with events measured across 7 quarters (21 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Harriet Lane Clinic, Baltimore, Maryland, United States